CLINICAL TRIAL: NCT00631826
Title: Shoulder Internal/External Rotational Flexibility is Related to Throwing Arm Injuries in Professional Baseball Players
Brief Title: Shoulder Rotational Flexibility and Throwing Arm Injuries of Baseball Pitchers
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Major League Baseball (Unknown)
Responsible Party: Sponsor
Other Study IDs: 50-2007
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Shoulder Injuries; Shoulder Flexibility; Rotational Resistance of Shoulder
Keywords: Shoulder; Injuries; Flexiblity; Rotational resistance
MeSH Terms: conditions — Shoulder Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The evaluation of any relationship between the rotational resistance of the shoulder and shoulder flexibility with throwing arm injuries in professional and college level pitchers.

ELIGIBILITY:
Inclusion Criteria:

* Currently competing
* Healthy pitching arm

Exclusion Criteria:

* Inactive status
* Previous injury

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Collegiate level baseball pitchers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Zheng, PhD, Principal Investigator — UF Department of Orthopaedics and Rehabilitation
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States